CLINICAL TRIAL: NCT01578174
Title: The Effect of Dexmedetomidine in the Management of Pain After Uterine Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Clinical assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2011-0928
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pain Control
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline 0.9%
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine(Dexmedetomidine 2 mL and normal saline 98 mL mixed -> 2㎍/mL) : the infusion of 0.2㎍/kg/hr is started at 30 minutes before the procedure and the infusion dose is raised to 0.4㎍/kg/hr after completion of procedure
  Arms: Dexmedetomidine
Drug: Normal saline 0.9% — Normal saline 100mL(guess as 2㎍/mL):the infusion of 0.2㎍/kg/hr is started at 30 minutes before the procedure and the infusion dose is raised to 0.4㎍/kg/hr after completion of procedure
  Arms: Control

SUMMARY:
The investigators examined the effect of dexmedetomidine in the management of pain after uterine artery embolization.

DETAILED DESCRIPTION:
Leiomyoma are the most common female reproductive tract tumors. Uterine artery embolization(UAE) is a minimally invasive treatment alternative to hysterectomy and myomectomy. However, post-procedural pain control after UAE remains a major problem. Therefore, the aim of study is to evaluate the efficacy of dexmedetomidine in pain control after UAE.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20,
* ASA class I and II

Exclusion Criteria:

* bradycardia (< 45 bpm)
* heart block
* liver failure
* renal failure
* uncontrolled hypertension
* body mass index ≥ 30 kg/m2

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption by patient-controlled analgesia | 24 hours

SECONDARY OUTCOMES:
Side effects | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea